CLINICAL TRIAL: NCT06372782
Title: A Randomized, Split-Hand, Subject-Blinded Study Comparing Pain, Safety and Effectiveness of Restylane Skinboosters Vital Lidocaine and Restylane Vital Without Lidocaine for Improved Appearance of the Dorsal Hand in Chinese Subjects
Brief Title: Comparing Pain, Safety and Effectiveness of Restylane Skinboosters Vital Lido and Vital Without Lido in Dorsal Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 43CH2305
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2024-03

CONDITIONS: Skin Aging of Dorsal Hands

STUDY DESIGN:
Who Masked: Participant
Masking Description: Each subject will receive treatment on Day 1 with Restylane Skinboosters Vital Lidocaine® in one hand and Restylane Vital in the opposite hand, as randomly assigned. Subject was kept bline is that he/she does not know which product treatment their hands received separately
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Skinboosters Vital Lidocaine (Experimental): Participant's one hand treated by Restylane Skinboosters Vital Lidocaine
  Interventions: Device: Restylane Skinboosters Vital Lidocaine
- Restylane Vital (Active Comparator): Participant's another hand treated by Restylane Vital
  Interventions: Device: Restylane Vital

INTERVENTIONS:
Device: Restylane Skinboosters Vital Lidocaine — Each subject will receive treatment on Day 1 with Restylane Skinboosters Vital Lidocaine in one hand and Restylane Vital in the opposite hand, as randomly assigned.
  Arms: Restylane Skinboosters Vital Lidocaine
Device: Restylane Vital — Each subject will receive treatment on Day 1 with Restylane Vital in one hand and the experimental device in the opposite hand, as randomly assigned
  Arms: Restylane Vital

SUMMARY:
This is a randomized, multi-center, split-hand, subject-blinded study comparing pain, safety and effectiveness of Restylane Skinboosters Vital Lidocaine and Restylane Vital without lidocaine for improving appearance of the dorsal hands in Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent to participate in the study
2. Chinese origin
3. Age at least 18 years
4. The subject is willing and able to comply with the requirements of the study and agrees to adhere to the visit schedule and to be compliant to the study instructions
5. Subjects eligible for treatment to improve appearance of the dorsal hand by increasing tissue volume
6. Same grade of tissue degeneration and need for treatment in both hands

Exclusion Criteria:

1. Any previous non-permanent or permanent implant/filler in the hands, including autologous fat
2. Any mesotherapy or resurfacing procedure (laser, chemical peels or other ablative or non-ablative treatment) in the hands within 6 months prior to baseline
3. Any previous hand surgery including sclerotherapy
4. Any fibrosis or scarring or deformities on the hands
5. Advanced photoaged/ photodamaged skin (e.g. advanced skin elastosis, multiple lentigo solaris lesions) or skin condition with very crinkled or fragile skin on the dorsal hands
6. Subjects with active skin disease, inflammation or related conditions in the hand
7. Subjects with a history of precancerous (e.g. actinic keratosis) or cancerous lesions in the hands
8. Subjects with a history of Raynaud´s disease or phenomenon, or history of other disease that may affect peripheral circulation
9. History of neurological disease that may affect peripheral neurological function
10. Subjects with a history of autoimmune disease or joint disease or connective tissue disease (e.g. rheumatoid arthritis, lupus, scleroderma etc)
11. Subjects with known hypersensitivity to any ingredient of the study product or anesthesia used in the study or with a history of any significant Adverse Events caused by dermal fillers
12. Use of topical retinoids on the dorsal hands within 6 weeks prior to baseline or use of systemic retinoids within 6 months prior to baseline
13. History of chronic lymph edema or breast cancer /mastectomy with potential to cause edema
14. Concomitant thrombolytic or anticoagulant therapy and therapy with inhibitors of platelet aggregation, (e.g. non-steriod anti-inflammatory drugs, acetylsalicylic acid, Omega 3 and Vitamin E) within 2 weeks prior to treatment, or a history of bleeding disorders. Cyclooxygenase-2 (COX-2) inhibitors are allowed
15. Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic or topical (dorsal hands) corticosteroids (inhaled corticoids are allowed) within three months before study treatment
16. History of untreated epilepsy or other significant medical conditions
17. Women who are pregnant or breast feeding, or Woman of childbearing potential who are not practicing adequate contraception or planning to become pregnant during the study period.
18. Subjects participating in another interventional clinical study within 30 days of baseline
19. Subjects with unattainable expectation with regard to the aesthetic results of the treatment
20. Subjects who are involved in conducting the study (e.g. colleagues within the same department) or close relatives to any of the study staffs (e.g. parents, children, siblings or spouse ) as well as subjects who are employed by the Sponsor company, or close relatives of employees at the Sponsor company
21. Subjects with any other condition which in the opinion of the Investigator, might compromise the subject's ability to tolerate the injection procedure or comply with requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galderma R&D, Study Director — Galderma R&D
Locations (3):
- China (3):
  - Galderma Research Site 01, Shanghai, Shanghai Municipality
  - Galderma Research Site 02, Hangzhou, Zhejiang
  - Galderma Research Site 03, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 90 participants were enrolled in this study, each participant received Restylane Skinbooster vital lidocaine treatment on one hand, and Restylane Vital on his/her other hand.
Units Other Than Participants: Hands
Groups:
- All Study Participants: Each subject received treatment on Day 1 with Restylane Skinboosters Vital Lidocaine in one hand and Restylane Vital in the opposite hand, as randomly assigned.
Period: Overall Study
Arm/Group | All Study Participants
Started | 90; 180 Hands
Restylane Skinboosters Vital Lidocaine-treated Hand | 90; 90 Hands
Restylane Vital-treated Hand | 90; 90 Hands
Completed | 90; 180 Hands
Not Completed | 0; 0 Hands

BASELINE CHARACTERISTICS:
Groups:
- Restylane Skinboosters Vital Lidocaine and Restylane Vital: Subjects' hands treated by Restylane Skinboosters Vital Lidocaine and Restylane Vital
  Each subject will receive treatment on Day 1 with Restylane Skinboosters Vital Lidocaine in one hand and Restylane Vital in the opposite hand, as randomly assigned.
Arm/Group | Restylane Skinboosters Vital Lidocaine and Restylane Vital
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 89
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 40.2 [22 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese Origin | 90
Region of Enrollment [Number; unit: participants]
  China | 90

OUTCOME MEASURES:

1. Primary Outcome: The Within-subject Difference in VAS Score (Restylane Skinboosters Vital Lidocaine- Restylane Vital) at End of Injection (T0).
Description: The VAS is a subjective scale to measure pain intensity. Total range is 0-100, 0 represents no pain and 100 represents the worst pain you can imagine, meaning a lower value is considered a better outcome in terms of a less painful treatment. The subject shall be instructed to put a vertical mark, approximating the pain experienced after the procedure, on a 100 mm horizontal line labelled "no pain" at the left end and "the worst pain you can imagine" at the right end. The distance in mm from the left end (no pain) to the subject's VAS mark shall be measured with a standard ruler. Each hand will be evaluated independently.
Time Frame: End of Injection (T0)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Restylane Skinboosters Vital Lidocaine: Subject's one hand treated by Restylane Skinboosters Vital Lidocaine
  Each subject will receive treatment on Day 1 with Restylane Skinboosters Vital Lidocaine in one hand.
- Restylane Vital: Subject's one hand treated by Restylane Vital.
  Each subject will receive treatment on Day 1 with Restylane Vital Lidocaine in another hand.
Arm/Group | Restylane Skinboosters Vital Lidocaine | Restylane Vital
Number analyzed (Participants) | 90 | 90
score on a scale | 32.5 (19.41) | 46.9 (23.43)
Statistical Analysis 1: Comparison: Restylane Skinboosters Vital Lidocaine vs Restylane Vital; Within-Subject Difference in VAS Score at the End of Injection (FAS); Test type: Superiority; p < 0.0001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Through study completion, up to 1 month.
Arm/Group | Restylane Skinboosters Vital Lidocaine and Restylane Vital
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 3/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Skinboosters Vital Lidocaine and Restylane Vital (N=90)
Conjunctival deposit (Eye disorders) | 1 (1)
Asthenia (General disorders) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT06372782/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT06372782/SAP_001.pdf